CLINICAL TRIAL: NCT00650715
Title: Effect of Acute and Chronic Whole-Body Vibration Exercise on Serum Insulin-Like Growth Factor-1 Levels in Women With Fibromyalgia
Brief Title: Effects of Whole-Body Vibration Exercise on Serum IGF-1 in Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Nacional d'Educacio Fisica de Catalunya (Other)
Responsible Party: Eduard Alentorn-Geli, MD, INEFC
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WBVIGF1FM
Record Dates: First submitted 2008-03-31; First posted 2008-04-02 (Estimated); Last update posted 2008-04-02 (Estimated); Status verified 2008-03

CONDITIONS: Fibromyalgia; Hormonal Responses to Exercise in Patients With Fibromyalgia.
Keywords: Fibromyalgia; Whole-Body vibration; Exercise; IGF-1
MeSH Terms: conditions — Fibromyalgia; Motor Activity

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- VG (Active Comparator): Vibration Group (VG) underwent a protocol with whole-body vibration exercise twice a week for a total of six weeks. The group continued with their usual pharmacological treatment.
  Interventions: Device: Vibratory platform, PowerPlate®, Badhoevendorp, Netherlands
- CG (Placebo Comparator): The Control Group (CG) underwent the same protocol of exercises than VG but without vibratory stimulus. The CG continued with their usual pharmacological treatment.
  Interventions: Device: Placebo Whole-body vibration exercise

INTERVENTIONS:
Device: Vibratory platform, PowerPlate®, Badhoevendorp, Netherlands — Six exercises (static and dynamic tasks) while standing on a Whole-body vibration platform. The six exercises (30 seconds each) were repeated six times with a recovery of 3 minutes in between. The Whole-body vibration intensity was kept constant at 30 Hz of frequency and 2 mm of amplitude.
  Arms: VG
Device: Placebo Whole-body vibration exercise — Six exercises (static and dynamic tasks) while standing on a Whole-body vibration platform. The six exercises (30 seconds each) were repeated six times with a recovery of 3 minutes in between. All exercises were performed without the influence of a vibratory stimulus.
  Arms: CG

SUMMARY:
The purpose of this study was to investigate the acute and chronic effect of whole-body vibration exercise on serum insulin-like growth factor-1 levels in women with fibromyalgia (FM). It was hypothesized that women with FM would exhibit an increase in IGF-1 following both acute and chronic WBV. Twenty-four women with FM were randomized into two groups: Vibration Group (VG) and Control Group (CG). The VG underwent a protocol with WBV exercise twice a week for a total of six weeks, whereas the CG performed the same protocol without vibratory stimulus. Both groups continued with their usual pharmacological treatment. Serum IGF-1 levels were determined using Enzyme-Linked Immunosorbent Assay (ELISA). To test the effect of chronic WBV, serum IGF-1 measurements were taken at baseline and at weeks 1,3, and 6 of intervention. To test the effect of acute WBV, within week 1, serum IGF-1 measurements were taken before and immediately following a session of WBV.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed of fibromyalgia according to the American College of Rheumatology criteria for at least three years.

Exclusion Criteria:

* Orthopedic limitation, or cardiovascular, pulmonary, or metabolic disease that would preclude exercise.
* Participation in any other study.

Ages: 35 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-12; Primary Completion 2005-01 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
Serum IGF-1 levels | Baseline, Week 1, Week 3, Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Eduard Alentorn-Geli, MD, Principal Investigator — INEFC
Locations (1):
- Institut Nacional d'Educación Física de Catalunya, Barcelona, Barcelona, Spain